CLINICAL TRIAL: NCT00067756
Title: "4 Phenyl Butyrate Mediated Secretion Rescue in Alpha 1-Antitrypsin Deficient Individuals"
Brief Title: 4-PBA: Will it Increase the Level of Alpha 1-Antitrypsin(AAT) in Persons With AAT Deficiency?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Alpha-1 Foundation (Other); Brantly, Mark L., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 87-2001
Record Dates: First submitted 2003-08-26; First posted 2003-08-27 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-04

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: Pulmonary Disease; Liver Disease
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Lung Diseases; Liver Diseases | interventions — 4-phenylbutylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 4-PBA (Experimental): The study will involve a 4-PBA dose escalation and pharmacokinetics component The study group will be comprised of a total of at least 10 AAT-deficient,(phenotype ZZ referred to as PiZZ) patients. These patients will be divided into two groups: with and without clinical evidence of mild to moderate hepatocellular injury.
  Interventions: Drug: 4-PBA

INTERVENTIONS:
Drug: 4-PBA — During the first 3 days of this phase baseline serum AAT levels will be determined. The participants will be then given increased amounts of 4-PBA orally in 6 divided doses (day 4-6, 30 g/day and day 7-9, 40/day
  Other Names: 4-phenyl butyric acid

SUMMARY:
The purpose of this study is to find out whether 4-PBA will increase the level of AAT in persons with AAT deficiency whether or not they have liver disease.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether 4-PBA will significantly increase serum Z AAT levels in AAT-deficient individuals with and without evidence of hepatocellular injury and to assess its effects on liver injury.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Serum A1-PI levels <11uM an appropriate genetic phenotype/genotype
* 5 of 10 subjects must have documented laboratory evidence of liver disease
* Willingness to withhold Prolastin therapy for 6 weeks prior to screening and throughout the 4-PBA dosing period (up to 3 months)

Exclusion Criteria:

* Any cause of liver disease other than Alpha-1 Antitrypsin deficiency
* Evidence of advanced liver disease
* HIV positive
* Use of systemic steroids, ursodeoxycholic acid (Actigall, Urso), or herbs in the prior 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2001-11; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
To determine if 4-PBA significantly increases secretion of AAT in AAT-deficient individuals with and without liver disease. | 10 days

SECONDARY OUTCOMES:
To determine the pharmacokinetics of 4-PBA | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Brantly, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Gonzalez-Peralta RP, Leonard S, Harvey R, Schreck P, Vironosvkaya N, Brantly ML. 4-PHENYL BUTYRATE MEDIATED SECRETION RESCUE IN PATIENTS WITH ALPHA 1-ANTITRYPSIN (AAT) DEFICIENCY: A PILOT STUDY HEPATOLOGY, Vol. 44, No. 4, Suppl. 1, 2006 AASLD ABSTRACTS, p. 211A, 61
- See also: Alpha-1 Foundation Alpha-1 Research Program — http://www.alphaone.ufl.edu